CLINICAL TRIAL: NCT03605810
Title: An Estimated Glomerular Filtration Rate (eGFR) Level Prediction
Brief Title: Study to Develop a Tool to Estimate the Kidney Function in Databases Without Laboratory Data
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20325
Record Dates: First submitted 2018-07-23; First posted 2018-07-30 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Renal Function
Keywords: Renal function, eGRF, Atrial fibrillation, Coronary artery disease, Type 2 diabetes mellitus, Machine learning, Prognostic modeling
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- eGFR-population: To be included in the eGFR-population, patients have to have at least one recorded eGFR value in the OPTUM CDM database between January 1, 2007 and December 31, 2016, be adults (>18 years of age at the time of eGFR test) and have at least 370/180 days (180 days serves as sensitivity analysis) of continuous enrollment in medical and pharmacy insurance plans since eGFR test date.
  Interventions: Other: No Intervention
- Atrial fibrillation (AF) sub-population: To be included in the AF sub-population patients need to satisfy the inclusion criteria for the eGFR-population; have two inpatient or outpatient diagnoses for AF or atrial flutter on two different days within the study period irrespective of time points when eGFR is measured.
  Patients with at least one inpatient or outpatient diagnosis or procedure code for mitral stenosis and prosthetic valves within the study period will be excluded.
  Interventions: Other: No Intervention
- Coronary artery disease (CAD) sub-population: To be included in the CAD sub-population patients need to satisfy the inclusion criteria for the eGFR-population; have at least one inpatient CAD diagnosis within the study period irrespective of time points when eGFR is measured.
  Interventions: Other: No Intervention
- Type 2 diabetes mellitus (T2DM) sub-population: To be included in the T2DM sub-population patients need to satisfy the inclusion criteria for the eGFR-population; have at least two inpatient or outpatient diagnosis of T2DM on two different days within the study period irrespective of time points when eGFR is measured.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This study is the development of algorithms/models to predict eGFR values and/or classes for patients at certain time point based on entries in claims database (demographic characteristics, clinical diagnoses, procedures and drug treatments) for a general population and a variety of use-cases (AF, CAD, T2DM patients sub-populations).

SUMMARY:
Scientific analyses are frequently performed on e.g. health insurance databases to study the usage and effectiveness of drugs in real life.

Kidney function is known to have an influence on a patients disease development and/or drug levels in blood.

However, often direct measures for kidney function are not available in databases.

This study plans to develop tools to classify the renal function of patients, which helps scientists to identify patient cohorts (groups of patients sharing same characteristics) for scientific analyses.

DETAILED DESCRIPTION:
Renal impairment is a common comorbidity in patients with diverse main underlying diseases and a pathology accompanying increasing age. Renal function might be an important modifier of treatment effects.

Population-based administrative claims databases are increasingly used in large-scale comparative outcomes studies of drug treatments. However, claims databases often lack information on laboratory tests results limiting their usefulness in Real-World Evidence(RWE) research of patients with renal impairment.

There is a need to develop methods for identification of patients with renal dysfunction from healthcare administrative claims-based proxies.

The main objective of this study is the development of algorithms/models to predict eGFR values and/or classes for patients at certain time point based on entries in claims database (demographic characteristics, clinical diagnoses, procedures and drug treatments) for a general population and a variety of use-cases (atrial fibrillation, coronary artery disease, type 2 diabetes mellitus patients sub-populations). To achieve this, modern data-driven machine learning techniques will be applied to discover relationships between renal status, measured by eGFR, and longitudinal patient-level data.

Evaluation of models' performance (out of sample validation, benchmark test, performance differences between eGFR value prediction algorithms and classification models tailored for the pre-defined eGFR classes) will be done as well.

ELIGIBILITY:
To be included in the eGFR-population, patients have to have at least one recorded eGFR value in the OPTUM CDM database between January 1, 2007 and December 31, 2016, be adults (>18 years of age at the time of eGFR test) and have at least 370/180 days (180 days serves as sensitivity analysis) of continuous enrollment in medical and pharmacy insurance plans since eGFR test date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with at least one recorded eGFR value in the OPTUM CDM database between January 1, 2007 and December 31, 2016 will be included in the use-case 1 "eGFR population". Further cases refer to the sub-populations of the eGFR-population, namely
  * Atrial fibrillation (AF) sub-population;
  * Coronary artery disease (CAD) sub-population;
  * Type 2 diabetes mellitus (T2DM) sub-population.
Sampling Method: Non-Probability Sample
Enrollment: 5132200 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Performance of classification to predict eGFR | From eGRF values starting and lasting 180d + 370d
  For numeric models cross-validated performance is measured as correlation via r*2.
  Class based performances are measured as cross-validated sensitivities given pre-defined false discovery rates with following definition for positives and negatives:
  Observed eGFR class X:
  * positive: eGFR measured at begin of time frame is in class X
  * negative: eGFR measured at begin of time frame is not in class X
  Class predicted by model:
  * positive: eGFR predicted is class X
  * negative: eGFR predicted is not class X

CONTACTS AND LOCATIONS:
Locations (1):
- US OPTUM CDM database, Whippany, New Jersey, United States